CLINICAL TRIAL: NCT03695640
Title: The Effect of Magnesium Sulfate Added to Levobupivacaine in Continous Femoral Block on Analgesic Requirements Following Total Knee Arthroplasty
Brief Title: Effect of Magnesium Sulphate on Analgesia Following Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Baturay Kansu Kazbek, Principle Investigator, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MgTKA
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Knee Arthroplasty, Total; Postoperative Pain
Keywords: total knee arthroplasty; postoperative pain; continuous femoral nerve block; magnesium sulphate
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Active Comparator): continuous femoral nerve block with levobupivacaine
  Interventions: Procedure: continuous femoral nerve block
- Group LM (Experimental): continuous femoral nerve block with levobupivacaine and magnesium sulfate
  Interventions: Drug: Magnesium Sulfate; Procedure: continuous femoral nerve block

INTERVENTIONS:
Drug: Magnesium Sulfate — Addition of magnesium sulfate as an adjuvant to levobupivacaine
  Arms: Group LM
Procedure: continuous femoral nerve block — continuous nerve block with levobupivacaine for treatment postoperative pain

SUMMARY:
This study is designed to investigate the effect of magnesium sulfate added to levobupivacaine in continuous femoral nerve block following total knee arthroplasty.

DETAILED DESCRIPTION:
Pain after knee arthroplasty is a serious concern. This study was designed to investigate the effect of magnesium sulfate added to levobupivacaine in continuous femoral nerve block on analgesic requirements following total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective unilateral primary total knee arthroplasty

Exclusion Criteria:

* Patient refusal to enroll in the study
* Patient refusal of neuraxial anesthesia
* Existence of contraindications for neuraxial anesthesia
* Known history of allergy to any of the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | T0:(Baseline) Postoperative 1st hour, T1: Change in 2nd, T2: Change in 4th, T3: Change in 6th, T4: Change in 12th, T5: Change in 24th, T6: Change in 36th, T7: Change in 48th, T8: Change in 72nd hours
  measurement of postoperative pain using Visual Analogue Score. Minimum: 0 Maximum: 10. Higher values represent more pain, hence lower values are better

SECONDARY OUTCOMES:
Analgesic consumption | T0:(Baseline) Postoperative 1st hour, T1: Change in 2nd, T2: Change in 4th, T3: Change in 6th, T4: Change in 12th, T5: Change in 24th, T6: Change in 36th, T7: Change in 48th, T8: Change in 72nd hours
  Consumption of local anesthetic in patient controlled analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Baturay K Kazbek, MD, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University Faculty of Medicine Hospital, Ankara, Balgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrecht E, Morfey D, Chan V, Gandhi R, Koshkin A, Chin KJ, Robinson S, Frascarolo P, Brull R. Single-injection or continuous femoral nerve block for total knee arthroplasty? Clin Orthop Relat Res. 2014 May;472(5):1384-93. doi: 10.1007/s11999-013-3192-3. PMID 23928707